CLINICAL TRIAL: NCT03730948
Title: Pilot Study of Mature Dendritic Cell Vaccination for Resected Hypermutated Colorectal Cancer
Brief Title: DC Vaccine in Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Pennsylvania (Other)
Collaborators: Parker Institute for Cancer Immunotherapy (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 16218, 831453; R01CA204261 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; cancer vaccine; dendritic cell vaccine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): All subjects will receive the vaccine and be followed per the schedule of procedures.
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — DC vaccine for colorectal cancer

SUMMARY:
This is a pilot study to assess the safety and tolerability, as well as the immune response rate, of mDC3 vaccine in patients with colorectal cancer.

DETAILED DESCRIPTION:
This is a pilot study to assess the safety and tolerability, as well as the immune response rate, of mDC3 vaccine in patients with colorectal cancer.

Eligible patients that provide written informed consent will undergo apheresis to collect blood mononuclear cells for vaccine production approximately 1 week prior to vaccine infusion. Each study subject will receive cyclophosphamide 300mg/m^2 intravenously 3 to 4 days prior to the vaccine dose to deplete regulatory T cells. For each vaccine dose, all subjects will receive autologous dendritic cells pulsed with mutated peptides. On Day 1, the subject will receive the primer vaccine dose; this will be followed by one booster vaccine dose approximately 8 weeks later. Peripheral blood will be taken weekly, and a second apheresis procedure will be performed at the end of study to monitor the immune response to the vaccine. Information will be gathered from usual clinic visits for approximately 1 year following the End of Treatment Study Visit to evaluate for disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed stage I and II hypermutated colorectal cancer (CRC)
* Surgically resected disease
* Male or female patients 18+ years of age
* ECOG performance status 0-1
* Certain laboratory values, performed within 14 days prior to consent
* Subjects of reproductive potential must agree to use a medically accepted birth control method during the trial and for at least two months following the trial.
* Provide written informed consent

Exclusion Criteria:

* Prior malignancy within 3 years that may put subject at risk
* Pregnant or nursing women
* Concurrent treatment with systemic immunosuppressants including corticosteroids, calcineurin inhibitors, antiproliferative agents within 2 weeks of consent. Local (inhaled or topical) steroids or replacement dose prednisone are permitted.
* Known allergy to eggs
* Any uncontrolled intercurrent illness or active ongoing infection thta may put subject at additional risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Reiss-Binder, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All subjects will receive the DC vaccine for colorectal cancer and be followed per the schedule of procedures. Each subject's vaccine is created using a panel of subject-specific (unique) tumor neoantigen peptides. Therefore, antigens tested for each subject are different.
  DC Vaccine #1: protocol-specified dose of 7.50x10^6 - 1.50x10^7 DC per peptide; minimum acceptable dose for infusion is 1.0x10^6 DC per peptide.
  DC Vaccine #2 and #3: 1.0x10^6 - 5.0x10^6 DC per peptide; minimum acceptable dose for infusion is 1.0x10^6 DC per peptide.
Period: Overall Study
Arm/Group | All Subjects
Started | 4
Completed | 2
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Changes in Numbers of Peptide-specific CD8+ T Cells (Post-vaccine Immune Response)
Description: Assessment of cellular immune activity may occur via the application of flow cytometry. Numbers of peptide-specific CD8+ T cells will be measured by flow cytometric-based intracellular cytokine or tetramer staining. Flow cytometric assays will include an examination of the influence of immunotherapy on the ability of subject T cells to exhibit phenotypic markers associated with cytolytic potential (e.g. IFN-y, IL-2, TNF-alpha, Granzyme B) after short-term stimulation by mutated peptide and p-HLA multimer staining. PBMC responses against a pool of known antigenic Cytomegalovirus, Epstein Barr Virus and Influenza epitopes will be evaluated in order to track general cellular immune competence during the study.
Time Frame: Screening, Day 1, Day 43, Day 85. Also at following timepoints, which will vary by subject: 7-14 days after last vaccine; 30 days after last vaccine; every 3 months beginning 6 months since first vaccine until month 12.
Population: Results are reported as IFN-G producing cells / 5x10^5 cells, all CD3+ T cells. Neither subject was tested at 6 months, 9 months, or 12 months time points.
Measure: Number; unit: IFN-G producing cells / 5x10^5 cells
Groups:
- Subject 01, Antigen TBCC1D23 K632X; Subject 01, Antigen CDC7 L28X; Subject 01, Antigen MSH3 K381X; Subject 01, Antigen NKTR 613-614X; Subject 01, Antigen DDX51 P492L; Subject 01, Antigen APC A885X; Subject 01, Antigen TCERG1 R889X; Subject 01, Antigen MAP3K21 A767V; Subject 01, Antigen DAG1 W31R; Subject 01, Antigen ZC3H18 A886V; Subject 01, Antigen PRR11 K20X; Subject 01, Antigen MSH6 Q657H; Subject 02, Antigen DOCK3 T1850X; Subject 02, Antigen FAM214BA42X; Subject 02, Antigen FHDC1F100X; Subject 02, Antigen DOCK1E1616X; Subject 02, Antigen PLA2G6 S359L; Subject 02, Antigen POLG2K160E; Subject 02, Antigen LYSMD3 V111A; Subject 02, Antigen FARR459H; Subject 02, Antigen PDHXI190L; Subject 02, Antigen FNIP2 K575E; Subject 02, Antigen ARID1AG284X; Subject 02, Antigen ACVR2AK435X: All subjects will receive the DC vaccine for colorectal cancer and be followed per the schedule of procedures. Each subject's vaccine is created using a panel of subject-specific (unique) tumor neoantigen peptides. Therefore, antigens tested for each subject are different.
Arm/Group | Subject 01, Antigen TBCC1D23 K632X | Subject 01, Antigen CDC7 L28X | Subject 01, Antigen MSH3 K381X | Subject 01, Antigen NKTR 613-614X | Subject 01, Antigen DDX51 P492L | Subject 01, Antigen APC A885X | Subject 01, Antigen TCERG1 R889X | Subject 01, Antigen MAP3K21 A767V | Subject 01, Antigen DAG1 W31R | Subject 01, Antigen ZC3H18 A886V | Subject 01, Antigen PRR11 K20X | Subject 01, Antigen MSH6 Q657H | Subject 02, Antigen DOCK3 T1850X | Subject 02, Antigen FAM214BA42X | Subject 02, Antigen FHDC1F100X | Subject 02, Antigen DOCK1E1616X | Subject 02, Antigen PLA2G6 S359L | Subject 02, Antigen POLG2K160E | Subject 02, Antigen LYSMD3 V111A | Subject 02, Antigen FARR459H | Subject 02, Antigen PDHXI190L | Subject 02, Antigen FNIP2 K575E | Subject 02, Antigen ARID1AG284X | Subject 02, Antigen ACVR2AK435X
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
IFN-G producing cells / 5x10^5 cells
  Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 0 | 1 | 33 | 0 | 27 | 36 | 0 | 0 | 0 | 1339 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 9 | 0 | 15 | 9
  Day 43 (week 6) | 201 | 0 | 234 | 312 | 65 | 240 | 0 | 0 | 0 | 650 | 5 | 17 | 5 | 0 | 43 | 0 | 34 | 0 | 0 | 0 | 289 | 75 | 0 | 618
  Day 85 (week 12) | 0 | 0 | 253 | 167 | 55 | 280 | 0 | 0 | 85 | 331 | 10 | 0 | 12 | 0 | 5 | 8 | 5 | 0 | 38 | 8 | 500 | 255 | 0 | 237
  7-14 days after last vaccine (week 14) | 53 | 0 | 286 | 13 | 306 | 352 | 0 | 0 | 9 | 432 | 10 | 3 | 5 | 4 | 19 | 10 | 5 | 2 | 2 | 29 | 414 | 491 | 0 | 80
  30 days after last vaccine | 325 | 0 | 1159 | 0 | 461 | 697 | 0 | 34 | 43 | 1250 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 789 | 453 | 20 | 2

2. Primary Outcome: Adverse Events Experienced by Subjects (i.e. Safety of DC Vaccine in Subjects With Surgically Resected Hypermutated CRC)
Description: Number of subjects who experienced adverse events. Detailed adverse event data is presented in the AE section.
Time Frame: Through study completion (at 12 months)
Population: The number of participants includes 1 subject who began the study but did not complete it.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 3
participants | 3

3. Secondary Outcome: Percentage of CD8+ Cells in Primary Tumor Tissue
Description: Descriptive models
Time Frame: as for outcome 1
Population: Per protocol, tissue samples will be used if obtained as part of standard of care procedures only. No samples were collected as part of standard of care procedures, therefore no analysis could be performed.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion (at 12 months)
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=4)
Nausea (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (3)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03730948/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03730948/ICF_001.pdf